CLINICAL TRIAL: NCT02255487
Title: A Phase IV, Multicenter, Prospective, Randomized, Controlled Clinical Study to Compare the Irrisept System Versus Standard of Care (SoC) on the Prevalence of Surgical Site Infections in Patients With Abdominal Trauma or Acute Surgical Abdomen
Brief Title: Irrisept Versus Standard of Care in the Prevention of Surgical Site Infections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated early after the Interim Analysis due, in part, to issues with the accuracy and completeness of the data collected.
Sponsor: Irrimax Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRR-CT-901-2013-01
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Results first posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: The randomization methodology was controlled by the site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- IrriSept System (Experimental): IrriSept device used for surgical irrigation in subjects with abdominal trauma or acute surgical abdomen
  Interventions: Device: IrriSept System
- Standard of Care (SoC) only (Active Comparator): Institution will provide routine Standard of Care (SoC) surgical preparation for subjects with abdominal trauma or acute surgical abdomen.
  Interventions: Other: No Intervention - Standard of Care (SoC) only

INTERVENTIONS:
Device: IrriSept System — The IrriSept system consists of two containers: Step1, a sterile bottle of 450 mL 0.05% Chlorhexidine Gluconate in 99.95% water and Step 2, a sterile bottle of 450 mL of sterile 0.9% Normal Saline. Step 1 and Step 2 are identical in shape and size, with a clear distinction in labeling between. Their unique design allows the solutions to be delivered under the ideal pressure as determined by the surgeon via manual compression for wound and surgical irrigation.
  Subjects randomized to the IrriSept system will receive irrigation per the provided Instructions for use; those randomized to Standard of Care will receive routine care per discretion of the investigator and in accordance with the institution's guidelines, which may or may not include some other type of irrigation.
  Arms: IrriSept System
Other: No Intervention - Standard of Care (SoC) only — Institution will provide routine Standard of Care (SoC) as surgical preparation for subjects with abdominal trauma or acute surgical abdomen.
  Arms: Standard of Care (SoC) only

SUMMARY:
The purpose of this study was to compare the rate of surgical site infections in patients randomized to Irrisept versus SoC, who had an open abdominal laparotomy for abdominal trauma or acute surgical abdomen.

DETAILED DESCRIPTION:
The trial was explained to potential subjects, the informed consent was completed and and eligibility was verified. After this, the subjects were randomized to Irrisept or SoC and an open abdominal laparotomy with primary closure due to (1) blunt or penetrating abdominal trauma or (2) acute surgical abdomen was performed. The follow-up visit was performed approximately 30 days later.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female, 18 years of age or older
2. Has provided written informed consent or has surrogate consent provided by a Legally Authorized Representative (LAR)
3. Has experienced abdominal trauma, blunt or penetrating, requiring open abdominal laparotomy with primary closure or
4. Has experienced acute surgical abdomen requiring open abdominal laparotomy with primary closure

Exclusion Criteria:

1. Known allergy to Chlorhexidine Gluconate (CHG)
2. Estimated Abbreviated Injury Scale (AIS) score of six (6) at the time of surgery, for all trauma patients
3. American Society of Anesthesiologists Physical Status Classification (ASA) score of five (5) or greater (As ASA scoring is a subjective measure, if the PI finds the patient stable enough for study participation despite a score of 5, enrollment may continue.)
4. Female volunteers who are pregnant and/or breast feeding
5. Damage control laparotomy
6. Abdominal incision created prior to operating room (i.e. incision made in trauma bay to cross clamp the aorta)
7. Currently enrolled in an ongoing, interventional, randomized clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Fry, MD, Study Director — Michael Pine Associates
Locations (17):
- United States (17):
  - The University of Arizona, Tucson, Arizona
  - The University of Southern California, USC Medical Center, Los Angeles, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - The University of South Florida, Tampa General Hospital, Tampa, Florida
  - The University of Iowa, Iowa City, Iowa
  - The University of Kentucky Research Foundation, Lexington, Kentucky
  - The University of Maryland, Baltimore, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Saint Louis University, St Louis, Missouri
  - The University of Cincinnati Health, Cincinnati, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - Regional One Health Research Institute, Memphis, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - The University of Washington, Harborview Medical Center, Seattle, Washington
  - The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2015 to 2017, patients with abdominal trauma or acute surgical abdomen were recruited from participating research sites' universities, hospitals and/or emergency departments.
Pre-assignment Details: The planned sample size was 1100 screened, 650 completed & 600 evaluated. However, the study was terminated early after the interim analysis due, in part, to issues with the accuracy and completeness of the data collected. There were 627 consented and 617 randomized subjects. The intent-to-treat (ITT) population was defined as all randomized subjects. Of these, 309 were randomized to Irrisept and 308 to Standard of Care.
Groups:
- Irrisept: For subjects randomized to the investigational group, Irrisept was used during the surgical procedure, per the provided instructions for use.
  Irrisept consists of two containers: (1) a sterile bottle of 450 mL of 0.05% Chlorhexidine Gluconate (CHG) in 99.95% sterile water and (2) a sterile bottle of 450 mL of sterile 0.9% normal saline.
- Standard of Care (SoC): For subjects randomized to the control group, any Standard of Care (SoC) irrigation solution, preferred by the site, was used during the surgical procedure.
Period: Overall Study
Arm/Group | Irrisept | Standard of Care (SoC)
Started | 309 | 308
Modified Intent to Treat (mITT) | 293 (Within the ITT population, subjects with unknown age entries (modified ITT or mITT) were considered "non-evaluable" and excluded from the analysis. The mITT population was defined as patients 18 years of age or older.) | 291 (Within the ITT population, subjects with unknown age entries (modified ITT or mITT) were considered "non-evaluable" and excluded from the analysis. The mITT population was defined as patients 18 years of age or older.)
Completed | 218 | 230
Not Completed | 91 | 78

BASELINE CHARACTERISTICS:
Groups:
- Irrisept: For subjects randomized to the investigational group, Irrisept was used during the surgical procedure, per the provided instructions for use.
- Standard of Care (SoC): For subjects randomized to the control group, any SoC irrigation solution, preferred by the site, was used during the surgical procedure.
- Total: Total of all reporting groups
Arm/Group | Irrisept | Standard of Care (SoC) | Total
Number analyzed (Participants) | 293 | 291 | 584
Age, Customized [Mean (Standard Deviation); unit: years]
  Average Age (Years) | 49.1 (18.7) | 50.1 (17.1) | 49.6 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 121 | 224
  Male | 190 | 170 | 360
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 199 | 202 | 401
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 8 | 3 | 11
  Black or African American | 75 | 77 | 152
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  Mixed Race | 0 | 1 | 1
  Other | 5 | 2 | 7
  Unknown | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 293 | 291 | 584
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29.0 (10.9) | 29.3 (12.2) | 29.2 (11.6)
Number of Participants By Surgical Case Type [Count of Participants; unit: Participants]
  Acute Surgical Abdomen | 180 | 191 | 371
  Trauma | 108 | 98 | 206
  Missing | 5 | 2 | 7
Average Height [Mean (Standard Deviation); unit: cm] | 172.7 (19.0) | 170.0 (14.4) | 171.4 (16.7)
Average Weight [Mean (Standard Deviation); unit: kg] | 85.2 (27.3) | 83.4 (25.8) | 84.3 (26.6)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With Surgical Site Infections (SSI)
Description: The primary endpoint was the rate of SSIs observed 30 days from the date of the index operation.
Time Frame: 30 (+/- 3) days post-surgical procedure
Population: Data is from the percentage of subjects that reported an SSI for the mITT subject populations.
Measure: Count of Participants; unit: Participants
Arm/Group | Irrisept | Standard of Care (SoC)
Number analyzed (Participants) | 293 | 291
Participants | 48 | 32

2. Secondary Outcome: Hospital Readmission Rates
Description: A secondary endpoint was the rate of Irrisept versus SoC subjects that required hospital readmission due to SSIs.
Time Frame: 30 (+/- 3) days post-surgical procedure
Population: Data is from the percentage of subjects that reported hospital readmission, due to an SSI, for the mITT subject populations.
Measure: Count of Participants; unit: Participants
Arm/Group | Irrisept | Standard of Care (SoC)
Number analyzed (Participants) | 293 | 291
Participants | 13 | 13

3. Secondary Outcome: Hospital Costs
Description: A secondary endpoint was the estimated hospital cost to charge ratio between Irrisept and SoC subjects. No data was collected towards this objective; thus, the success or failure of this endpoint was not assessed.
Time Frame: 0 days
Population: No data was collected for either randomization group, towards this objective. Therefore, the success or failure of this endpoint was not assessed.
Arm/Group | Irrisept | Standard of Care (SoC)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Length of Hospital Stay
Description: A secondary endpoint was the length of hospital stay between subjects randomized to Irrisept versus SoC.
Time Frame: 30 (+/- 3) days post-surgical procedure
Population: Data is from the average number of days in the hospital for the mITT subject populations.
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Irrisept | Standard of Care (SoC)
Number analyzed (Participants) | 293 | 291
number of days | 11.6 (24.8) | 12.0 (23.4)

ADVERSE EVENTS:
Time Frame: Adverse events were not collected.
Description: Adverse events were not collected.
Arm/Group | Irrisept | Standard of Care (SoC)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT02255487/Prot_SAP_000.pdf